CLINICAL TRIAL: NCT05922124
Title: Cefiderocol and Ampicillin-sulbactam vs. Colistin or Colistin-meropenem for Carbapenem Resistant Acinetobacter Baumannii Bacteremia or Hospital-acquired Pneumonia: Controlled Clinical Study With Historical Controls (CASCADE)
Brief Title: Cefiderocol and Ampicillin-sulbactam vs. Colistin +/- Meropenem for Carbapenem Resistant A. Baumannii
Acronym: CASCADE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Monaldi Hospital (Other); Rutgers Robert Wood Johnson Medical School (Other); Pisa University Hospital (Unknown); Assaf-Harofeh Medical Center (Other Government); Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V0.1 May 2023
Record Dates: First submitted 2023-05-31; First posted 2023-06-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Carbapenem Resistant Bacterial Infection; Acinetobacter Bacteremia; Acinetobacter Pneumonia
MeSH Terms: interventions — Cefiderocol; sultamicillin; Colistin; Meropenem

STUDY DESIGN:
Intervention Model Description: Controlled clinical study with historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cefiderocol + ampicillin-sulbactam (Experimental): Cefiderocol 2 gram intravenous (IV) q8 hours and ampicillin-sulbactam 3 gram IV q6 hours for patients with normal creatinine clearance, both administered as extended infusion of 3 hours. Dosing adjusted according to reduced and augmented renal clearance and to renal replacement therapies.
  Interventions: Drug: Cefiderocol; Drug: Ampicillin-sulbactam
- Colistin or colistin + meropenem (Active Comparator): Colistin 9 million units (MIU) intravenous (IV) loading dose followed by 4.5 MIU for patients with normal creatinine clearance +/- meropenem 2 gram IV administered as extended infusion of 3 hours. Dosing adjusted according to reduced and augmented renal clearance and to renal replacement therapies.
  Interventions: Drug: Colistin; Drug: Meropenem

INTERVENTIONS:
Drug: Cefiderocol — Test drug regimen
  Other Names: Fetroja
  Arms: Cefiderocol + ampicillin-sulbactam
Drug: Ampicillin-sulbactam — Synergistic combination
  Other Names: Unasyn
  Arms: Cefiderocol + ampicillin-sulbactam
Drug: Colistin — Historical comparator
  Arms: Colistin or colistin + meropenem
Drug: Meropenem — Historical comparator synergistic combination
  Arms: Colistin or colistin + meropenem

SUMMARY:
Patients with bloodstream infections, hospital acquired pneumonia or ventilator-associated pneumonia caused by carbapenem-resistant Acinetobacter baumannii (CRAB) treated with cefiderocol combined with ampicillin sulbactam will be compared to patients treated treated with colistin alone or colistin combined with meropenem.

DETAILED DESCRIPTION:
This will be a prospective controlled clinical study with historical controls.

In the prospective CASCADE study consecutive consenting patients with bloodstream infections, hospital acquired pneumonia or ventilator-associated pneumonia will be treated with cefiderocol combined with ampicillin sulbactam in 3 hospitals in Israel and 2 hospitals in Italy, all endemic for CRAB. We plan to recruit 150 patients into this prospective studies.

The CASCADE cohort will be compared to patients treated for the same types of infection in two recently completed randomized controlled trials (AIDA and OVERCOME). These trials compared between treatment with colistin vs. treatment with colistin-meropenem combination therapy, both finding no difference between treatment groups among patients with carbapenem-resistant Acinetobacter baumannii (CRAB) pneumonia. Thus, patients in CASCADE will be compared to all patients with CRAB bloodstream infections, hospital acquired pneumonia or ventilator-associated pneumonia in these randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

Adults >18 years with bacteremia or hospital-acquired pneumonia (HAP)/ ventilator-associated pneumonia (VAP) (Table 3) caused by carbapenem-resistant A. baumannii (CRAB) (meropenem and/ or imipenem minimal inhibitory concentration (MIC) >8 μg/mL) susceptible to cefiderocol (disc zone diameter >=17 mm, corresponding to an MIC <2 μg/mL). We will include CRAB regardless of colistin, ampicillin-sulbactam, minocycline, tigecycline, trimethoprim/sulfamethoxazole and/or aminoglycoside susceptibility of the isolate. Attribution of the HAP/ VAP to CRAB will be allowed with isolation of CRAB from any respiratory sample within 7 days prior to the clinical diagnosis of pneumonia.

Exclusion Criteria:

* More than 72 hours of therapy with in-vitro coverage against the CRAB within 96 hours of enrolment
* Polymicrobial carbapenem-susceptible infections: growth of other pathogens susceptible to carbapenems, or another beta-lactam, deemed clinically-significant by the treating physicians in blood or sputum (with HAP/ VAP). We will allow recruitment of patients with other carbapenem-resistant Gram-negative bacteria
* CRAB susceptible any beta-lactam other than cefiderocol
* Coronavirus 2019 (COVID-19) co-infection
* Immediate-type hypersensitivity to penicillin
* Pregnant women
* Previous participation in the trial
* Lack of informed consent, considering the procedures acceptable to ethics committees per locale, including deferred consent
* Infection requiring treatment for over 14 days, at the discretion of the investigators
* Life expectancy less than 24 hours or expected futility of antibiotic treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 734 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 28 days
  Death from any cause

SECONDARY OUTCOMES:
All cause mortality | 14 days
  Death from any cause
Clinical failure | Day 10-14
  Composite of:
  * Death
  * Systolic blood pressure ≤90 mmHg or need for vasopressor support
  * Worsening sequential organ failure assessment score (SOFA) score, define as:
    * for baseline SOFA ≥ 3: stable or increased
    * for baseline SOFA <3: any increase
  * For patients with hospital-acquired pneumonia (HAP)/ ventilator-associated pneumonia (VAP), partial pressure of oxygen in arterial blood (PaO2)/ fraction of inspired oxygen (FiO2) ratio worsened
  * For patients with bacteremia, growth of the initial isolate in blood cultures after ≥ 5 days since study treatment start
Microbiological failure | Day 5-7
  Isolation of the initial isolate (phenotypically identical) in blood cultures 5 days or more after start of treatment or in respiratory samples 7 days or more.
Resistance development to cefiderocol | 28 days
  Development of carbapenemase-producing Enterobacterales (CPE), non-CPE carbapenem-resistant Enterobacterales (CRE), carbapenem-resistant A. baumannii (CRAB) and carbapenem-resistant Pseudomonas aeruginosa (CRPA) resistance to cefiderocol in clinical and surveillance cultures collected as defined in the study's protocol
Hospital stay | 28 days
  Among 28-day survivors
Decline in functional capacity | 28 days
  Functional capacity will be assessed in four categories: independent; requires some assistance; requires assistance for activities of daily living (ADL); and bedridden. Decline in functional capacity will be defined as any 1-category worsening.
Adverse event - Clostridiodes difficile infection | 28 days
  Diarrhea with a positive C. difficile toxin test
Adverse event - renal failure | 28 days
  Renal failure due to any reason using the RIFLE ( risk, injury, failure, loss, End stage kidney disease) criteria (classifying patients to None, Risk, Injury, Failure, Loss and ESRD) at day 14 and day 28 and defined as worsening by two RIFLE categories (e.g. from Risk to Failure, etc.)
Adverse event - Acute liver injury | 28 days
  Increase in aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3-fold or increased bilirubin >2 above upper limits of normal (ULN) or baseline value if higher than ULN.

OTHER OUTCOMES:
Desirability of Outcome Ranking (DOOR) | 28 days
  Defined DOOR outcome analysis: Alive no event; Alive 1 event; Alive 2 events; Alive 3 events; Dead. The DOOR events will be: (1) Clinical failure as defined above (2) Hospital stay >14 days from enrolment (3) Adverse events: renal failure, Clostridiodes difficile infection or acute liver injury

CONTACTS AND LOCATIONS:
Overall Officials: Marco Falcone, Principal Investigator — Pisa University Hospital; Dafna Yahav, Principal Investigator — Sheba Medical Center; Mical Paul, Principal Investigator — Rambam Health Care Campus
Locations (3):
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Sheba Tel HaShomer Medical Campus, Ramat Gan
  - Shamir Medical Center (Assaf Harofeh), Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be published. At the end of the study the database will be made available from the lead author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As soon as published
Access Criteria: Justification to lead author

REFERENCES:
- [Background] Paul M, Daikos GL, Durante-Mangoni E, Yahav D, Carmeli Y, Benattar YD, Skiada A, Andini R, Eliakim-Raz N, Nutman A, Zusman O, Antoniadou A, Pafundi PC, Adler A, Dickstein Y, Pavleas I, Zampino R, Daitch V, Bitterman R, Zayyad H, Koppel F, Levi I, Babich T, Friberg LE, Mouton JW, Theuretzbacher U, Leibovici L. Colistin alone versus colistin plus meropenem for treatment of severe infections caused by carbapenem-resistant Gram-negative bacteria: an open-label, randomised controlled trial. Lancet Infect Dis. 2018 Apr;18(4):391-400. doi: 10.1016/S1473-3099(18)30099-9. Epub 2018 Feb 16. PMID 29456043
- [Background] Kaye KS, Marchaim D, Thamlikitkul V, Carmeli Y, Chiu CH, Daikos G, Dhar S, Durante-Mangoni E, Gikas A, Kotanidou A, Paul M, Roilides E, Rybak M, Samarkos M, Sims M, Tancheva D, Tsiodras S, Kett D, Patel G, Calfee D, Leibovici L, Power L, Munoz-Price S, Stevenson K, Susick L, Latack K, Daniel J, Chiou C, Divine GW, Ghazyaran V, Pogue JM. Colistin Monotherapy versus Combination Therapy for Carbapenem-Resistant Organisms. NEJM Evid. 2023 Jan;2(1):10.1056/evidoa2200131. doi: 10.1056/evidoa2200131. Epub 2022 Dec 6. PMID 37538951